CLINICAL TRIAL: NCT02252887
Title: Phase II Study of Gemcitabine, Trastuzumab, and Pertuzumab in the Treatment of Metastatic HER2-Positive Breast Cancer After Prior Trastuzumab/Pertuzumab- or Pertuzumab-Based Therapy
Brief Title: Gemcitabine, Trastuzumab, and Pertuzumab in the Treatment of Metastatic HER2-Positive Breast Cancer After Prior Trastuzumab/Pertuzumab, or Pertuzumab Based Therapy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: Genentech, Inc. (Industry); Hoffmann-La Roche (Industry); Hartford HealthCare (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 14-124
Record Dates: First submitted 2014-09-26; First posted 2014-09-30 (Estimated); Last update posted 2025-07-25 (Actual); Status verified 2025-07

CONDITIONS: Metastatic HER2-Positive Breast Cancer
Keywords: Gemcitabine,; Trastuzumab; Pertuzumab; 14-124
MeSH Terms: interventions — Gemcitabine; Trastuzumab; pertuzumab

ARMS (1):
- Gemcitabine, Trastuzumab, and Pertuzuma (Experimental): The regimen will consist of gemcitabine at 1000mg/m^2 IV weekly days 1 + 8 q 3 weeks + trastuzumab every 3 weeks (8 mg/kg loading dose followed by 6 mg/kg every 3 weeks) + pertuzumab every 3 weeks (840 mg as a loading dose followed by 420 mg every 3 weeks), all given intravenously (IV). Trastuzumab may be given IV weekly (4 mg/kg loading dose followed by 2 mg/kg weekly) in lieu of the every 3 week schedule. A loading dose of trastuzumab will not be required for patients who have received it < 6 weeks prior to Cycle 1 Day 1.
  Interventions: Drug: Gemcitabine; Drug: Trastuzumab; Drug: Pertuzumab

INTERVENTIONS:
Drug: Gemcitabine
Drug: Trastuzumab
Drug: Pertuzumab

SUMMARY:
The purpose of this study is to see if a combination of drugs can help to treat breast cancer. This is a Phase II study which will test whether this combination of drugs is effective and will provide further information on side effects and safety. A standard chemotherapy, gemcitabine, will be combined with 2 other drugs that target the HER2 receptor. The HER2 receptor is a growth protein on the surface of some breast cancer cells that provides messages telling the breast cancer cell to grow. The standard chemotherapy will be gemcitabine.. The other two drugs work against HER2. One is called trastuzumab (Herceptin) and it is commonly given to women with advanced and early HER2 positive breast cancer. The other drug, pertuzumab (Perjeta), is also given to women with advanced HER2 positive breast cancer. The drugs in this study are each individually approved for the treatment of metastatic breast cancer. However, this study is looking at the effectiveness of gemcitabine with trastuzumab and pertuzumab when given to women who have advanced HER2 positive breast cancer who have had prior trastuzumab + pertuzumab or pertuzumab-based therapy.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ to 18
* Stage IV HER2 (+) breast cancer
* Histologically documented HER2 (+) breast cancer as defined as IHC 3+ or FISH amplification of ≥ 2.0 of primary or metastatic site; results from the local lab are acceptable.
* lECOG performance status 0 -1
* Prior treatment with trastuzumab + pertuzumab (HP)-based therapy or pertuzumab-based in the neoadjuvantadjuvant, unresectable, locally advanced, or metastatic setting.
* ≤ 3 prior chemotherapies in the metastatic setting. Prior anthracycline, taxane, gemcitabine, and anti-HER2 agents (i.e. trastuzumab, pertuzumab, lapatinib, neratinib, TDM-1, etc.) are allowed. If patients received prior gemcitabine, it could not have been combined with pertuzumab. Patients should have progression of disease on current therapy.
* Measurable or non-measurable disease.
* LVEF ≥ 50%
* Hematologic parameters: white blood cell (WBC) count of ≥ 3000/ul, absolute neutrophil count (ANC) ≥ 1000/ul, platelets ≥ 100,000/ul, hemoglobin ≥10.0 g/dl
* Non-hematologic parameters: bilirubin ≤ 1.5 mg/dl, AST/ALT≤ 2.5 x upper limit of normal (ULN), alkaline phosphatase ≤ 5 x ULN.
* Creatinine ≤ 1.5 mg/dl
* Patients with "treated and stable" brain lesions of a duration of ≥ 2 months may be enrolled.

Exclusion Criteria:

* History of prior unstable angina, myocardial infarction, CHF, uncontrolled ventricular arrhythmias within 12 months
* History of prior ≥ G 3 hypersensitivity (HSR) or any toxicity to trastuzumab or pertuzumab that warranted permanent cessation of this agent
* History of hepatitis B or C
* Pregnant patients

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2015-01-12 (Actual); Primary Completion 2025-07-24 (Actual); Study Completion 2025-07-24 (Actual)

PRIMARY OUTCOMES:
progression free | 3 months
  Progression-free survival (PFS) is defined from time from treatment assignment to disease progression or death, whichever comes first. The primary endpoint is PFS and secondary endpoint will include the response rate using the RECIST criteria (version 1.1).

SECONDARY OUTCOMES:
progression-free survival | 2 years
  Progression-free survival (PFS) is defined from time from treatment assignment to disease progression or death, whichever comes first.
response | 2 years
  Response to treatment will be determined using both RECIST and PRC ( PET Response Criteria criteria).
overall survival | 2 years
  Progression-free survival and median overall survival will also be estimated by the Kaplan-Meier method.
safety | 2 years
  This study will use the NCI Common Toxicity Criteria (CTC) AE version 4.0 for toxicity.

CONTACTS AND LOCATIONS:
Overall Officials: Chau Dang, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (5):
- United States (5):
  - Hartford Healthcare Cancer Institute @ Hartford Hospital, Hartford, Connecticut
  - Memorial Sloan Kettering at Basking Ridge, Basking Ridge, New Jersey
  - Memorial Sloan Kettering Monmouth, Middletown, New Jersey
  - Memorial Sloan Kettering Westchester, Harrison, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York

REFERENCES:
- [Derived] Iyengar NM, Smyth LM, Lake D, Gucalp A, Singh JC, Traina TA, DeFusco P, Fornier MN, Goldfarb S, Jhaveri K, Modi S, Troso-Sandoval T, Patil S, Ulaner GA, Jochelson M, Norton L, Hudis CA, Dang CT. Efficacy and Safety of Gemcitabine With Trastuzumab and Pertuzumab After Prior Pertuzumab-Based Therapy Among Patients With Human Epidermal Growth Factor Receptor 2-Positive Metastatic Breast Cancer: A Phase 2 Clinical Trial. JAMA Netw Open. 2019 Nov 1;2(11):e1916211. doi: 10.1001/jamanetworkopen.2019.16211. PMID 31774522
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org/